CLINICAL TRIAL: NCT00537186
Title: A Non-Comparative Open-Label Study of Iron Oligosaccharide in CHF Patients With Iron Deficiency (Either Absolute or Functional) Anaemia and a Need for Parenteral Iron
Brief Title: A Study of Iron Oligosaccharide in CHF Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-CHF-01; EudraCT No.: 2007-000764-25
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Heart Failure, Congestive
Keywords: Congestive heart failure; Anaemia; Iron oligosaccharide
MeSH Terms: conditions — Heart Failure; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Iron oligosaccharide
  Interventions: Drug: Iron oligosaccharide

INTERVENTIONS:
Drug: Iron oligosaccharide
  Other Names: MonoFer

SUMMARY:
The purpose of this study is to determine the safety profile of iron oligosaccharide in patients with congestive heart failure with a need for parenteral iron.

DETAILED DESCRIPTION:
Iron dextrans have been marketed for more than 50 years and the compiled preclinical and clinical experience with iron dextrans in general is well established. Pharmacosmos A/S already markets the iron dextran CosmoFer® worldwide, except in the US where the product is named INFeD®. A new iron oligosaccharide has been manufactured by Pharmacosmos A/S and it is a further development of CosmoFer® where ferric hydroxide has been combined with low molecular weight oligosaccharides in a relatively strong complex. This iron carbohydrate complex builds on the well established efficacy and safety profile of existing iron dextran but with a significantly reduced anaphylactic potential.

In order to ensure that iron oligosaccharide will not lead to unexpected adverse events the existing clinical information on iron dextrans in general needs to be supplied with clinical safety data from a limited number of relevant patients exposed to iron oligosaccharide in open label non-comparator studies.

The primary objective of the present study is to obtain safety reassurance with the use of iron oligosaccharide given either as repeated IV boluses or as total dose infusion for the correction of anaemia in patients with congestive heart failure in order to ensure that iron oligosaccharide will not lead to unexpected adverse events in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Congestive heart failure
* ≥ 18 years of age at screening
* Haemoglobin < 110 g/L (or 6.8 mmol/L)
* Serum ferritin < 800 µgram/L
* Life expectancy beyond 12 months
* Willingness to participate after written informed consent

Exclusion Criteria:

* Non iron deficiency anaemia
* Iron overload or disturbances in utilisation of iron (e.g. haemochromatosis, haemosiderosis)
* Drug hypersensitivity (i.e. previous hypersensitivity to iron dextran or iron mono- or disaccharide complexes)
* Patients with a history of multiple allergies
* Decompensated liver cirrhosis and hepatitis (alanine aminotransferase > 3 times normal) Acute or chronic infections Rheumatoid arthritis with symptoms or signs of active inflammation. Pregnancy and nursing. To avoid pregnancy, women have to be postmenopausal, surgically sterile, sexually inactive or practice reliable contraception Active bleeding Planned elective surgery during the study where significant blood loss is expected Participation in any other clinical trial within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Adverse events (AE) (Number and type of AE) | Eight weeks after enrollment
Serious adverse events (SAEs) | Eight weeks after enrollment
Physical examination | At screening visit and at end of study
Vital signs | At every visit
Clinical laboratory tests (biochemistry, haematology) | At every visit

SECONDARY OUTCOMES:
Change from baseline in haemoglobin, haematocrit, s-iron, transferrin saturation, and ferritin levels | At every visit

CONTACTS AND LOCATIONS:
Overall Officials: Per Hildebrandt, MD, Principal Investigator — Roskilde University Hospital, Medicinsk afdeling
Locations (1):
- Roskilde University Hospital, Medicinsk afdeling, Roskilde, Denmark